CLINICAL TRIAL: NCT00992069
Title: A Phase I, Safety, Tolerability, and Pharmacokinetic Interaction Study of Single-Dose TMC207 and Efavirenz in Healthy Volunteers
Brief Title: Safety, Tolerability, and Effect of TMC207 and Efavirenz in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5267; 10749 (Registry Identifier: DAIDS ES); ACTG A5267
Record Dates: First submitted 2009-10-01; First posted 2009-10-08 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis; HIV
Keywords: ARV; Pharmacokinetics; TMC207; Efavirenz
MeSH Terms: conditions — Tuberculosis | interventions — efavirenz; bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMC207 alone and with EFV (Experimental): Participants will receive single-dose TMC207 alone and then single-dose TMC207 with EFV.
  Interventions: Drug: Efavirenz (EFV); Drug: TMC207

INTERVENTIONS:
Drug: Efavirenz (EFV) — Oral dose of 600 mg daily, taken in the evening
  Other Names: Sustiva
Drug: TMC207 — Single oral dose of 400 mg in the morning

SUMMARY:
Common treatments for tuberculosis (TB) can interfere with certain antiretroviral (ARV) medications used to treat HIV. People whose immune systems are weakened by HIV infection are susceptible to TB, so it is important to find treatments for both that can be given in combination. This study will test the safety of combining a new medication for TB with an already approved HIV medication in healthy adults.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the second most deadly infectious disease after HIV. Multidrug-resistant TB (MDR-TB) has emerged as a worldwide epidemic, limiting treatment options. HIV infected people with suppressed immune systems are particularly susceptible to TB, and TB is the leading cause of death among people with HIV. Treating people infected with both HIV and TB is particularly problematic because rifamycins, the drug class usually used to treat TB, lower the effectiveness of certain anti-HIV medications. Studies of pharmacokinetics (PK), the interactions between drugs and body, are needed to determine which anti-TB and anti-HIV medications can be safely and effectively combined. This study will examine TMC207, a new anti-TB medication with the potential to shorten TB treatment time, combined with efavirenz (EFV), an antiretroviral (ARV) medication used in many first-line treatment regimens for HIV. The study will test PK and safety of this combination in healthy volunteers.

Participation in this study will last 49 days. At entry, participants will complete basic assessments, including taking a medical history and completing a physical exam, an eye exam, an electrocardiogram (ECG) to measure heartbeat, a pregnancy test, and a blood test. Certain behaviors and substances will be prohibited during the study, including consuming grapefruit, alcohol, or caffeine (on PK visit days); taking nutritional supplements, over-the-counter herbal medicines, and certain medicines and drugs from other studies; and excessive smoking. Participants will also be asked to keep a medication diary to record all medications they take during the study.

All participants will receive study medications on the same schedule: a single dose of TMC207 on Days 1 and 29, and daily dosing of EFV on Days 15 to 43.

Participants will complete two PK visits, one from Days 1 to 3, and one from Days 28 to 31. During PK visits, participants will have their vital signs checked and undergo an ECG, and they may also complete a limited physical exam, give a medication history, and report on symptoms. They will have multiple blood samples taken via a catheter left in place for the 3-day visit. Blood samples will be taken before receiving TMC207; 1, 2, 3, 4, 5, 6, 8, and 12 hours after receiving TMC207; and again on the mornings of Days 2 and 3.

Participants will complete six outpatient visits over the 11 days following each PK visit and one outpatient visit on Day 21, between PK visits. At outpatient visits participants will complete a blood draw and may complete a limited physical exam and medical history, record symptoms, and review their medication diaries.

On Day 49 participants will complete their last study visit, repeating many of the assessments from baseline testing. In the case of side effects or abnormal blood tests, participants may be monitored longer for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Females not of reproductive potential, defined as women who have been postmenopausal for at least 24 consecutive months or women who have undergone hysterectomy, bilateral oophorectomy, or bilateral tubal ligation
* Females who have been surgically sterilized and all males must agree to use contraceptives if participating in sexual activity that could lead to pregnancy while receiving the protocol-specified medications and for 4 weeks after stopping the medication
* Absence of HIV-1 infection, as documented by any licensed enzyme-linked immunosorbent assay (ELISA) test kit, within 21 days prior to study entry
* Estimated creatinine clearance of more than 50 ml/min, within 21 days prior to study entry, calculated by the Cockcroft-Gault method
* Laboratory test results obtained within 21 days prior to entry, including negative pregnancy test, negative hepatitis B and C tests, and certain blood values

Exclusion Criteria:

* Use of any prescription medication known to inhibit or induce CYP3A metabolizing enzymes within 30 days prior to entry
* Planned use during the study, from day 0 through the last PK blood draw, of any of the following: prescription medication(s), herbal supplement(s), nutritional supplement(s), or over-the-counter medication(s). Multivitamins and acetaminophen, up to 650 mg every 6 hours as an analgesic, are permitted.
* Hospitalization for any reason, pharmacotherapy for serious illness, or use of any prescription medication(s) within 14 days prior to study entry
* Receipt of any investigational study drug within 21 days prior to study entry
* Known allergy, sensitivity, or hypersensitivity to EFV or TMC207 or components of their formulations, including cyclodextrin allergy
* Significant previous or active history of cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease(s), as determined by the site investigator. This is inclusive of chronic illnesses or gastrointestinal conditions that may affect drug absorption, etc. Additionally, any medical condition that, in the opinion of the site investigator, would interfere with the volunteer's ability to participate in the protocol will exclude participation.
* Active illicit drug use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Suspicion of active tuberculosis (TB) by the site investigator
* Inability to abstain from alcoholic beverages, grapefruit, and grapefruit juice for the duration of the study
* For smokers, inability to smoke 5 cigarettes per day or less for the duration of the study
* Breastfeeding
* Electrocardiogram (ECG) showing first-degree or greater heart block or QT interval (QTc) greater than 440 ms within 21 days prior to study entry. First-degree heart block is defined as PR interval greater than 200 ms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) over 336 hours of TMC207, measured when dosed alone and when dosed together with efavirenz (EFV) 600 mg daily | Measured at baseline and Days 1 to 15, 28, and 29 to 43
Signs or symptoms of toxicity ranked Grade 2 or higher, according to the DAIDS adverse event (AE) grading table | Throughout study

SECONDARY OUTCOMES:
Maximum observed plasma or serum concentration (Cmax) and oral clearance (CL/F) of TMC207 and AUC, Cmax, and CL/F of the M2 metabolite of TMC207 when dosed alone and when dosed together with EFV 600 mg daily | Measured at baseline and Days 1 to 15, 28, and 29 to 43
AUC over 24 hours, Cmax, Cmin, CL/F, and elimination half-life (T1/2) of EFV and host EFV metabolism genotype status (CYP2B6) obtained from whole blood samples taken at screening | Measured at baseline and on Day 28
Correlation between AUC over 24 hours of EFV and AUC over 336 hours of TMC207 | Measured at baseline and Days 1 to 15, 28, and 29 to 43

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD, Study Chair — Johns Hopkins University
Locations (5):
- United States (5):
  - Ucsf Aids Crs, San Francisco, California
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Unc Aids Crs, Chapel Hill, North Carolina
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee

REFERENCES:
- [Background] Goldman RC, Plumley KV, Laughon BE. The evolution of extensively drug resistant tuberculosis (XDR-TB): history, status and issues for global control. Infect Disord Drug Targets. 2007 Jun;7(2):73-91. doi: 10.2174/187152607781001844. PMID 17970220
- [Background] McIlleron H, Meintjes G, Burman WJ, Maartens G. Complications of antiretroviral therapy in patients with tuberculosis: drug interactions, toxicity, and immune reconstitution inflammatory syndrome. J Infect Dis. 2007 Aug 15;196 Suppl 1:S63-75. doi: 10.1086/518655. PMID 17624828
- [Background] Diacon AH, Pym A, Grobusch M, Patientia R, Rustomjee R, Page-Shipp L, Pistorius C, Krause R, Bogoshi M, Churchyard G, Venter A, Allen J, Palomino JC, De Marez T, van Heeswijk RP, Lounis N, Meyvisch P, Verbeeck J, Parys W, de Beule K, Andries K, Mc Neeley DF. The diarylquinoline TMC207 for multidrug-resistant tuberculosis. N Engl J Med. 2009 Jun 4;360(23):2397-405. doi: 10.1056/NEJMoa0808427. PMID 19494215